CLINICAL TRIAL: NCT03356912
Title: CABAzitaxel With or Without Prednisone in Patients With Metastatic CAstration REsistant Prostate Cancer (mCRPC) Progressed During or After a Previous Docetaxel-based Chemotherapy:a Multi-center,Prospective,Two-arm, Open Label, Non Inferiority Phase II Study
Brief Title: CABAzitaxel With or Without Prednisone in Patients With Metastatic CAstration REsistant Prostate Cancer Progressed During or After a Previous Docetaxel-based Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: CABACARE
Record Dates: First submitted 2017-10-26; First posted 2017-11-29 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer; Castration-resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cabazitaxel plus prednisone (Active Comparator): Cabazitaxel 25 mg/m² intravenously (Day 1) every 3 weeks, plus prednisone 10 mg orally given daily. Premedication must be administered according to Cabazitaxel Package Insert.
  Interventions: Drug: Cabazitaxel; Drug: Prednisone
- Cabazitaxel (Experimental): Cabazitaxel 25 mg/m² intravenously (Day 1) every 3 weeks. Premedication must be administered according to Cabazitaxel Package Insert.
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel — Cabazitaxel drug products should be administered only by intravenous route.
  Prednison should be administered by oral route
Drug: Prednisone — Prednisone should be administred by oral route
  Arms: Cabazitaxel plus prednisone

SUMMARY:
Patients with metastatic castration resistant prostate cancer (mCRPC) progressed during or after a previous docetaxel-based chemotherapy, for whom cabazitaxel has been scheduled as per clinical practice and label indication.

In the "TROPIC" Trial, cabazitaxel, administered concomitantly with prednisone 10 mg daily, showed a significant advantage vs. mitoxantrone in both Overall Survival (OS) and Progression Free Survival (PFS) / radiographic PFS in patients failing docetaxel-based chemotherapy. Similar to docetaxel, cabazitaxel has been approved in combination with daily prednisone, but the benefits of adding daily corticosteroids to taxane chemotherapy remain to be proven. In fact, corticosteroids have a variety of biological effects, and a number of studies in large cohorts of patients show that they may have both favourable effects, mediated by adrenal androgen and cytokine suppression, and detrimental effects related to their adverse events associated with their long-term use as well to the potential promiscuous activation of the AR. In fact, prednisone and dexamethasone can activate some AR variants that make tumors sensitive to glucocorticoids even at low concentrations. It has been showed that point mutations of the AR, which appear to cluster in the ligand-binding domain, are rare in therapy naive patients but occur in 15- 45% of patients with castration-resistant disease and can increase AR affinity for a wide range of steroids. On the other hand, insofar as safety is concerned, omitting daily corticosteroids does not seem to increase toxicity (e.g. hypersensitivity reactions). In fact, in the CHARTEED trial, docetaxel was safely administered without daily corticosteroids. Safety data about the use of cabazitaxel without daily prednisone/prednisone alone are missing.

The CABACARE study is designed to assess the effects in terms of efficacy, safety as well as quality of life of omitting daily corticosteroids in patients treated with cabazitaxel. Furthermore, the CABACARE study evaluates the mutational status of the RB gene as well as presence of AR-V7 variant. The AR-V7 status assessed in circulating tumor cells has a strong predictive value for abiraterone/enzalutamide effectiveness, but its role in patients receiving cabazitaxel requires to be defined.

DETAILED DESCRIPTION:
Patients will be randomly assigned (1:1) to receive either:

Arm A Cabazitaxel 25 mg/m² intravenously (Day 1) every 3 weeks, plus prednisone 10 mg orally given daily. Premedication must be administered according to Cabazitaxel Package Insert.

Arm B Cabazitaxel 25 mg/m² intravenously (Day 1) every 3 weeks, without daily prednisone. Premedication must be administered according to Cabazitaxel Package Insert.

Each patient will be treated until radiological disease progression, unacceptable toxicity, or patient refusal. Patients will be followed through subsequent therapy lines of treatments until death or the study cut-off, whichever comes first.

Every effort will be made to administer the full dose regimen to maximize dose-intensity.

Dose reduction and/or treatment delay and/or treatment discontinuation are planned in case of severe toxicity. If toxicity occurs, dose of Cabazitaxel can be reduced to 20 mg/mq in both arms. If a second dose reduction is required the patient should be withdrawn from study.

Prednisone doses should not be delayed or modified or stopped (unless there is a contraindication to continue, the decision will be let to the investigator's discretion).

In case a dose reduction is required, cabazitaxel dose cannot be re-escalated. Prophylactic use of G-CSF is allowed, as per EORTC / ASCO guidelines and according to physician judgment. Patients experiencing neutropenia G 3-4 have to receive G-CSF in prophylaxis in subsequent cycles.

Primary Objective(s)

To evaluate whether cabazitaxel alone is non inferior in terms of radiographic PFS with respect to cabazitaxel plus daily prednisone in patients with castration resistant prostate cancer

Secondary Objective(s)

Safety in the two treatment arms; Health-Related Quality of Life (HRQL) and pain; Objective Response Rate (ORR) according to Response Evaluation Criteria In Solid Tumors (RECIST 1.1); Biochemical response (assessed considering PSA decrease ≥50% and waterfall plot results); Time to PSA Progression (TTPP); Radiographic Time to Progression (rTTP); Overall Survival (OS); Association of Overall

l Survival (OS), Progression Free Survival (PFS) and Objective Response Rate (ORR) with AR-V7 and RB status in circulating tumor cells assessed at flow-cytometry; Time to Skeletal-Related Event (SRE);

Primary end Point

Radiographic Progression-Free Survival (rPFS).

Secondary end points

Safety in the two treatment arms; Health-Related Quality of Life HRQL and pain; Objective Response Rate (ORR) according to Response Evaluation Criteria In Solid Tumors (RECIST 1.1); Biochemical response (PSA decrease ≥50%, waterfall plot); Time to PSA Progression (TTPP); Radiographic Time To Progression (rTTP); Overall Survival (OS); Association of Overall Survival (OS), Progression Free Survival (PFS) and Objective Response Rate (ORR) with AR-V7 and RB status in circulating tumor cells by the use of a DNA test; Time to Skeletal-Related Event (SRE).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Histological diagnosis of prostate adenocarcinoma;
3. Metastatic castration-resistant disease with documented radiographic progression (osseous or measurable lesions) during or after a docetaxel-based chemotherapy;
4. Testosterone level in the castration range (levels <50 ng/dl) because of a previous, and ongoing, androgen deprivation with LH-RH agonists or antagonists or bilateral orchiectomy;
5. Prior surgery and/or radiation therapy (to less or equal than 30% of the bone marrow) are allowed. However, at least 4 weeks must have been elapsed since surgery or completion of radiation therapy and the patient must has recovered from side effects;
6. Life expectancy ≥ 3 months;
7. Age > 18 years;
8. ECOG performance status 0-2;
9. ANC ≥ 1.5 x 109/L;
10. PLT ≥ 100 x 109/L;
11. Hb ≥ 10 g/dl;
12. Serum total bilirubin ≤ UNL;
13. AST/SGOT and/or ALT/SGPT ≤1,5 x ULN;
14. Serum Creatinine ≤1,5 times UNL (in case of limit values of serum creatinine, creatinine clearance calculated by CKD-EPI formula should be ≥60 ml/min);
15. PT or INR and PTT <1,5 times UNL (Note: patients who receive anti-coagulation treatment will be allowed to participate provided that any abnormality in these parameters exists);
16. Patients must be accessible for treatment and follow up;

Exclusion Criteria:

1. Participation in clinical trials with other investigational drug within 28 days of study entry;
2. Symptomatic or uncontrolled brain metastases. Patients with neurological symptoms must undergo a computed tomography (CT) scan/magnetic resonance imaging (MRI) of the brain to exclude brain metastasis; previously treated brain metastases will be allowed as long as the patient is neurologically stable and does not require steroids and anticonvulsants;
3. Less than 4 weeks elapsed from prior anticancer-therapy or surgery to the time of randomization. Prior treatment with abiraterone or enzalutamide is allowed and is used as a stratification factor at randomization. Patient may be on biphosphonates prior to study entry;
4. Less than 4 weeks from palliative Radiotherapy to time of randomization;
5. Any of the following within 6 months prior to study enrollment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, NYHA class III or IV congestive heart failure, stroke or transient ischemic attack, pulmonary embolism or other uncontrolled thromboembolic event;
6. Any severe acute or chronic medical condition which could impair the ability of the patient to participate to the study or interfere with interpretation of study results, or patient unable to comply with the study procedures;
7. Unstable diabetes mellitus, resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, acute diverticulitis or other contraindications to use of corticosteroid treatment;
8. Peripheral neuropathy Grade > 2 (National Cancer Institute Common Terminology Criteria (NCI CTCAE v.4.03);
9. Previous beta or gamma Isotope treatment (e.g. strontium or samarium), alpha emitters are allowed;
10. History of severe hypersensitivity reaction (> grade 2) to polysorbate 80 containing drugs;
11. Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a 2-week washout period is necessary for patients who are already on these treatments);
12. Previous malignancy except for basal cell or squamous cell skin cancer adequately treated, or any other cancer from which the patient has been disease-free for ≥ 5 years;
13. Patients with reproductive potential who do not agree to use accepted and effective method of contraception, based on the investigator's judgment, during the study treatment period.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-11-22 (Actual); Primary Completion 2021-05-04 (Estimated); Study Completion 2021-05-04 (Estimated)

PRIMARY OUTCOMES:
change from Baseline radiographic progression | From date of randomization until the date of first documented progression or but also during follow-up in case study treatment was discontinued without radiographic progression up to 48 months"
  Radiographic progression evaluated by RECIST 1.1 criteria with bone scan, chest abdominal and pelvi TC MRI

SECONDARY OUTCOMES:
Health-Related Quality of Life and pain | from the date of randomization and the date of either first documented pain progression or death due to any cause, whichever is earlier up to 48 months"
  Pain response will be calculated among patients with baseline median present pain intensity score (PPI) ≥2 on the McGill-Melzack scale and/or baseline mean analgesic score (AS) ≥10 points and with stable analgesia at baseline.
Adverse events | From date of randomization until the date of first documented progression or but also during follow-up in case study treatment was discontinued up to 48 months" "
  Incidence of Treatment-Emergent Adverse Events
Health-Related Quality of Life | From date of screening until the date of first documented progression up to 48 months"
  Functional Assessment of Cancer Therapy-Prostate" (FACT-P) questionnaire, version 4. The results is summed to give a score in the range of 0-156, where higher values represent better HRQL. Questionnaires will be self-administered and takes approximately 10 minutes to complete.
AR-V7 and RB status in circulating tumor cells | only at baseline
  genetic blood evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giuseppe, MD, Principal Investigator — Università Federico II Napoli
Locations (1):
- University Federico II of Naples, Naples, Italy